CLINICAL TRIAL: NCT00722332
Title: Evaluation of HepaGam B® in Combination With Antiviral Treatment in Hepatitis B Liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cangene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HB-009
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis B; Liver Transplantation
Keywords: HBIG (Hepatitis B Immune Globulin); Chronic Hepatitis B Recurrence; Liver Transplant
MeSH Terms: conditions — Hepatitis B | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HBV-related liver transplant patients
  Interventions: Biological: HepaGam B

INTERVENTIONS:
Biological: HepaGam B — Hepatitis B Immunoglobulin

SUMMARY:
The purpose of the study is to assess the pharmacokinetics, safety and efficacy of HepaGam B in combination with antiviral therapy for the prevention of hepatitis B virus (HBV) recurrence following HBV-related orthotopic liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* HBsAg-positive candidates for HBV-related liver transplant
* Treatment with antiviral therapy before transplantation as per treating physician's recommendation. (NOTE: It is expected that most patients will receive Lamivudine or Adefovir Dipivoxil pre-transplant. In the case of antiviral resistance, an effective alternative antiviral agent(s) must be used.)

Exclusion Criteria:

* Multi-organ transplantation recipients
* Liver re-transplantation except for primary non-function
* Presence of a hepatoma (larger than 5.0 cm as a solitary node) or 2 to 3 multi-focal nodes (larger than 3.0 cm each) (Milan Criteria) based on information available at baseline visit (CT scan, MRI).
* Patients requiring an OLT (Orthotopic Liver Transplant)due to fulminant hepatitis B
* OLT patients receiving a liver graft from a donor that is positive for HBsAg
* Patients using interferon pre-transplant (as interferon cannot be used post-transplant)
* History of IgA (immunoglobulin A) deficiency
* History of hypersensitivity to blood products.
* HIV or HCV positive
* Use of an investigational product, or participation in another clinical trial during the course of the study (with the exception of quality-of-life or repository studies)
* Pregnancy or planned pregnancy during the course of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of HepaGam B in combination with antiviral therapy | 15 month follow-up

SECONDARY OUTCOMES:
Pharmacokinetic profile and safety of HepaGam B in combination with antiviral therapy | 15 month follow-up

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - Los Angeles, California
  - Palo Alto, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Burlington, Massachusetts
  - Minneapolis, Minnesota
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
- Montreal, Quebec, Canada